CLINICAL TRIAL: NCT00050674
Title: Docetaxel and Gemcitabine With Filgrastim-SD/01 Support in Patients With Advanced Non-Small Cell Lung Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Schwartzberg, Lee, M.D. (Individual)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD01-20010120
Record Dates: First submitted 2002-12-17; First posted 2002-12-18 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer, oncology, neutropenia, chemotherapy, filgrastim
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms; Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Filgrastim-SD/01 (Experimental): 6 mg SC, Day 9, 24 hours after the end of the chemotherapy infusion
  Interventions: Drug: Filgrastim-SD/01

INTERVENTIONS:
Drug: Filgrastim-SD/01 — 6 mg SC on Day 9 (24 hours after the end of the chemotherapy infusion)

SUMMARY:
Determine whether patients have a decreased incidence of grade 3 and grade 4 neutropenia when Filgrastim-SD/01 is given with docetaxel and gemcitabine in patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Docetaxel and Gemcitabine given on day 1 and 8 of a 21-day schedule has substantial activity in non-small cell lung cancer. Both first and second-line patients have response rates comparable to or better than other standard combination regimens. Grade 3/4 neutropenia occurs in up to half of patients not given growth factor support.

Studies demonstrate that a single dose of Filgrastim-SF/01 at 100 mg/kg effectively enhances post chemotherapy neutrophil recovery in a manner similar to that of daily Filgrastim. This current study is designed to characterize the incidence of grade 3/4 neutropenia when a fixed dose of Filgrastim-SD/01 is added to a well-studied myelosuppressive chemotherapy regimen consisting of Gemcitabine and Docetaxel.

ELIGIBILITY:
* Histologically or cytologically documented non-small cell lung cancer
* Subjects must have stage IV or IIIB NSCLC
* 0-1 prior treatment regimens of chemotherapy
* Subjects must have bi-dimensionally measurable disease or evaluable disease by physical exam or radiological studies
* Age > 18 years
* 1st Line - ECOG 0-2
* 2nd Line - ECOG 0-1
* Absolute neutrophil count > or = 1.5 x 10 to the 9th power/L
* Platelet count > or = 100 x 10 to the 9th power/L
* Adequate renal function with screening serum creatinine < or = 2.0 mg/dL
* Adequate AST and ALT no more than 1.5 x the upper limit of normal and serum bilirubin < or = upper limit of normal
* Subjects must be at least two weeks from prior major thoracic or abdominal surgery and at least two weeks from completion of radiation therapy, and recovered from all toxicities associated with these treatments
* Negative HCG by urine or blood test in subject of child-bearing potential
* Life expectancy > 2 months
* Ethical - Before any study specific procedure is done or before study medication is administered, the subject or legally acceptable representative must give informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Schwartzberg, MD, FACP, Principal Investigator — The West Clinic, PC
Locations (2):
- United States (2):
  - The West Clinic, PC, Southaven, Mississippi
  - The West Clinic, PC, Memphis, Tennessee

REFERENCES:
- See also: Related Info — http://westclinic.com